CLINICAL TRIAL: NCT02875457
Title: A Randomized Controlled Study of Apatinib as the Maintenance Therapy for Extensive Stage Small Cell Lung Cancer After Combined With Etoposide and Cisplatin Chemotherapy
Brief Title: Apatinib as the Maintenance Therapy for Extensive Stage Small Cell Lung Cancer After Combined With Etoposide/Cisplatin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Dong Wang, chief physician, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEP-ES-SCLC
Record Dates: First submitted 2016-06-11; First posted 2016-08-23 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer; apatinib; etoposide; cisplatin
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Patients receive etoposide 100mg/m2 from day 1 to day 3, cisplatin 80mg/m2 on day 1, and apatinib 250mg/d , repeated every 21 days, a total of 6 cycles, and then continue to take apatinib 250mg/d until progressive Disease(PD).
  Interventions: Drug: apatinib;etoposide and cisplatin
- Arm B (Placebo Comparator): Patients receive etoposide 100mg/m2 from day 1 to day 3, cisplatin 80mg/m2 on day 1, and placebo, repeated every 21 days, a total of 6 cycles, and then continue to take placebo until PD.
  Interventions: Drug: placebo;etoposide and cisplatin

INTERVENTIONS:
Drug: apatinib;etoposide and cisplatin
  Arms: Arm A
Drug: placebo;etoposide and cisplatin
  Arms: Arm B

SUMMARY:
Apatinib has been approved as a second-line treatment for advanced gastric cancer. Several phase III clinical studies of non small cell lung cancer, liver cancer, colorectal cancer and other tumors also showed apatinib has less toxic side effects and better patient tolerance. However, the clinical application of apatinib in small cell lung cancer is still lack of evidence-based medicine. Etoposide and cisplatin chemotherapy is the first-line treatment for small-cell lung cancer. The purpose of this multicenter, randomized, prospective study is to investigate the efficacy and safety of apatinib as the maintenance therapy for extensive stage small cell lung cancer after combined with etoposide and cisplatin chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of small cell lung caner(SCLC), Extensive Stage.
* No prior cisplatin-based chemotherapy or radiotherapy.
* Males or females between 18 Years to 75 Years.
* Performance status of 0～2 on the ECOG criteria.
* Expected survival is above three months.
* At least one measurable lung tumor lesion (according to RECIST criteria, the application of conventional technology, diameter length of the lesion >= 20mm or spiral CT >=10mm).
* Adequate hematologic (Leukocyte count >= 4.0×109/L, neutrophil count>=2.0×109/L, hemoglobin>=95g/L, platelets>=100×109/L), hepatic function (aspartate transaminase (AST) & alanine transaminase(ALT) =<upper normal limit(UNL) x1.5, bilirubin level =< UNL x 1.5).
* Patient can take oral medicine.
* Patients have the ability to understand and voluntarily sign the informed consent, and allow adequate follow-up.

Exclusion Criteria:

* History of cardiovascular disease: congestive heart failure (CHF) > New York Heart Association (NYHA) II, active coronary artery disease(patients with myocardial infarction six months ago can be recruited), arrhythmias need to be treated (allow taking beta blockers or digoxin).
* Serious clinical infection (> NCI-CTCAE version 4.0 ,infection standard II).
* Patients with epilepsy who need to take medicine (such as steroids or anti epilepsy agents).
* with brain metastases.
* The patients had accepted allogeneic organ transplantation.
* Bleeding tendency or coagulation disorders.
* patients who need renal dialysis.
* suffered from other tumor within 5 years( Except: cervical carcinoma in situ, cured basal cell carcinoma, cured bladder epithelial tumor).
* uncontrolled hypertension (systolic pressure>150 mmHg , or diastolic pressure> 90 mmHg).
* thrombosis or embolism(cerebrovascular accidents including transient ischemic attack within the last 6 months).
* pulmonary hemorrhage >CTCAE grade 2 within 4 weeks before first use of drugs.
* Other organ hemorrhage >CTCAE grade 3 within 4 weeks before first use of drugs.
* severe uncured wounds, ulcers or fracture.
* uncured dehydration.
* Drugs abuse and medical, psychological or social conditions may interfere with the patient's participation in research or the results of the evaluation effect.
* Patients are allergic to drugs used in research.
* Factors influencing the safety and compliance of patients.
* Inability to comply with protocol or study procedures.
* Pregnant or breast-feeding.
* The researcher believe that the Patient is not suitable to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6 months
  The first day of treatment to the date that disease progression is reported.

SECONDARY OUTCOMES:
Overall survival | 5 years
  The first day of treatment to death or last survival confirm date.
Tumor response rate | 3 months
  The ratio between the number of responders and number of patients assessable for tumor response.
Treatment-related adverse events | the first date of treatment to 30 days after the last dose of study drug,assessed up to 6 months
  Treatment-related adverse events are assessed by common terminology criteria for adverse events(CTCAE) V4.0.
Performance Status | the first date of treatment to 30 days after the last dose of study drug, assessed up to 6 months
  Performance Status of patients will be assessed by Zubrod-Eastern cooperative oncology group(ECOG)-world health organization(WHO).

CONTACTS AND LOCATIONS:
Overall Officials: Wang Dong, PH.D., Principal Investigator — Daping Hospital, Third Military Medical University, Chongqing,China

IPD SHARING:
Plan to Share IPD: Undecided